CLINICAL TRIAL: NCT04422613
Title: Characterization of Persistent Pulmonary Abnormalities Following COVID-19 Pneumonia
Acronym: PULCO-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/20/0181
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Viral
Keywords: COVID-19; Respiratory Function Tests; Pulmonary Gas Exchange : Respiratory Tract Diseases; Pulmonary Embolism; Respiratory Distress Syndrome
MeSH Terms: conditions — Pneumonia, Viral; COVID-19; Pulmonary Embolism; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- characterization of pulmonary damage (Experimental): This clinical trial will be characterized the pulmonary damage after COVID-19 pneumonia
  Interventions: Diagnostic Test: pulmonary anomalies 4 months after documented COVID-19 pneumonia

INTERVENTIONS:
Diagnostic Test: pulmonary anomalies 4 months after documented COVID-19 pneumonia — Characterization of pulmonary damage with a complete pulmonary assessment 4 months after COVID-19 pneumonia,

SUMMARY:
Severe Acute Respiratory Syndrome (SARS) SARS-CoV-2, name of the Coronavirus Group of international Committee on taxonomy of viruses, is an emerging virus from the family of coronaviridae, responsible for the COVID-19 pandemic. This infection can progress to viral pneumonia, and in 3% of cases up to acute respiratory distress syndrome (ARDS) which conditions the prognosis of the disease.

Due to its unusual clinical presentation with a risk of sudden deterioration on the 8th day as a result of possible hyperinflammatory response, the respiratory impairment of COVID is unique and many questions remain unanswered concerning its evolution once the acute phase has passed. Knowledge of the evolution of pulmonary involvement, particularly in patients requiring hospitalization, can help reduce the morbidity linked to the persistent abnormalities identified by establishing early therapeutic management. It can also provide a better understanding of the mechanisms of pulmonary involvement in the acute phase. Current data regarding the acute phase of COVID-19 suggest that persistent abnormalities remain distant from this infection at all levels of the respiratory system: gas exchange, perfusion, ventilatory mechanics, and interstitial lung disease.

The main objective is to characterize persistent gas exchange anomalies 4 months after documented COVID-19 pneumonia, resulting in oxygen desaturation and requiring hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patient with COVID-19 pneumonia
* Positive PCR for COVID-19 on respiratory sample (saliva, nasopharyngeal, bronchial, tracheal aspiration or LBA)
* Having required hospitalization in the pulmonology service, intensive care in pneumology or resuscitation service at the Toulouse University Hospital
* Saturation <94% in ambient air at diagnosis
* Patient having a chest CT-scan proving pneumonia during his hospitalization
* Patient ≥ 18 years old
* Patient who has given written consent to participate in the study

Exclusion Criteria:

* Patient hospitalized for pneumonia not documented by a chest CT-scan
* Patient with negative COVID PCR
* Patient known before the episode of COVID-19 pneumonia for a respiratory or cardiac pathology which can lead in itself to an alteration of gas exchanges
* Patient under curators / guardianship
* Pregnant patient
* Minor patient
* Absence of consent for participation in the study
* Medical condition that does not allow for pulmonary function test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Alteration of the DLCO | 4 month
  Alteration of the DLCO test defined by a corrected DLCO value <70% of theoretical and / or desaturation in the 6 Minute Walk Test (loss of 4% or more of SpO2)

SECONDARY OUTCOMES:
Mechanism of the alteration of gas exchanges | 4 month
  The mechanism of the alteration of gas exchanges will be specified by the analysis of the values obtained during the diffusing CO / NO test, at 4 month after COVID- 19 pneumonia
Measurement on lung volumes | 4 month
  The mechanism of the alteration of gas exchanges will be specified by the analysis of the other values obtained during the measurement of lung volumes in respiratory function tests at 4 month after COVID- 19 pneumonia
mechanism of the alteration of gas exchanges by chest scan | 4 month
  The mechanism of the alteration of gas exchanges will be specified by the analysis of the other values obtained during chest CT-scan at 4 month after COVID- 19 pneumonia
mechanism of the alteration of gas exchanges by scintigraphy | 4 month
  The mechanism of the alteration of gas exchanges identified will be specified by the analysis of the other values obtained during pulmonary scintigraphy, at 4 month after COVID- 19 pneumonia :
Respiratory symptom | 4 month
  the existence of respiratory symptoms, defined by dyspnea, cough, sputum, haemoptysis, chest pain, sign of right ventricular failure, sleep disorders or a 6-minute walk test value <80% of theoretical, at 4 month after COVID- 19 pneumonia
Bronchial or ventilatory anomalies | 4 month
  the existence of persistent bronchial or ventilatory anomalies at 4 months, defined on current respiratory function tests (plethysmography, forced oscillometry test, diaphragmatic explorations, measurement of exhaled NO)
Persistent respiratory anomalies | 12 month
  Persistent respiratory anomalies at 4 months will be evaluated at 12 months of the acute episode by an appropriate paraclinical assessment : mechanism of the alteration of gas exchanges, Respiratory symptom and bronchial or ventilatory anomalies will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Elise Noël-Savina, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Noel-Savina E, Viatge T, Faviez G, Lepage B, Mhanna LT, Pontier S, Dupuis M, Collot S, Thomas P, Idoate Lacasia J, Crognier L, Bouharaoua S, Silva Sifontes S, Mazieres J, Prevot G, Didier A. Severe SARS-CoV-2 pneumonia: Clinical, functional and imaging outcomes at 4 months. Respir Med Res. 2021 Nov;80:100822. doi: 10.1016/j.resmer.2021.100822. Epub 2021 Apr 28. PMID 34242974